CLINICAL TRIAL: NCT05310201
Title: Targeting Teacher Stress and Well-being to Improve Child Outcomes: Impact of the Be Well Care Well Program
Brief Title: Impact of the Be Well Care Well Program on Early Care Education Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Delaware (Other); National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00105341; U54GM104941 (NIH)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Burnout, Caregiver
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Be Well Care Well (Experimental)
  Interventions: Behavioral: Be Well Care Well
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Be Well Care Well — Be Well Care Well addresses teacher well-being through activities implemented in the classroom aimed at reducing teacher stress and improving physical activity. A subset of teachers involved in the program will complete classroom observations and cortisol testing to examine additional measures of stress.
  Arms: Be Well Care Well

SUMMARY:
The study will address the following specific aims: (1) assess the impact of the BWCW program on teacher stress and physical activity, (2) Examine feasibility of collecting cortisol.

ELIGIBILITY:
Inclusion Criteria:

Teachers that meet the following criteria will be included:

1. currently employed as a teacher or assistant teacher at a participating ECE center;
2. ages 18 or older;
3. men or women;
4. able to speak, read, and write English.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC Department of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Teacher attention toward well-being as usual.
Period: Overall Study
Arm/Group | Be Well Care Well | Control
Started | 115 | 67
Completed | 71 | 45
Not Completed | 44 | 22

BASELINE CHARACTERISTICS:
Population: No different from assignment.
Groups:
- Control: Teacher well-being addressed as usual
- Total: Total of all reporting groups
Arm/Group | Be Well Care Well | Control | Total
Number analyzed (Participants) | 115 | 67 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 115 | 67 | 182
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13) | 40 (13.2) | 38.75 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 67 | 182
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 51 | 136
  White | 30 | 16 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 115 | 67 | 182

OUTCOME MEASURES:

1. Primary Outcome: Change in Score of Child Worker Job Stress Inventory
Description: The Child Worker Job Stress Inventory is a survey used to measure job stress via questionnaire that the childcare worker completes. This survey measure contains 22 items that range from 22 (low levels of stress) to 110 (High Levels of Stress). A higher score on each item represents higher child worker stress. The total score is utilized in this study with higher total score representing higher reported child worker job stress.
Time Frame: Baseline and 1 year follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Be Well Care Well: The Be Well Care well group includes those who received the Be Well Care Well Intervention.
- Control: The control group included the centers that did not receive the intervention (Be Well Care Well).
Arm/Group | Be Well Care Well | Control
Number analyzed (Participants) | 115 | 67
units on a scale | 25.1 (13.4) | 32.8 (21.4)

2. Primary Outcome: Change in Score on the Devereux Adult Resilience Survey
Description: The Devereux Adult Resilience Survey (DARS) is a 23-item self-report measure assessing personal strengths and resilience. Each item is scored from 0 (Not Yet) to 2 (Almost Always), yielding a raw total score range of 0-46. In this study, subscale scores (e.g., relationships, internal beliefs, professional skills) may be combined or analyzed separately. If a composite score is used, the method of combination (e.g., summing across subscales) will be specified in the analysis plan.
Time Frame: Baseline and 1-year follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Social networks, internalized beliefs, and resilience reported as usual in the daycare centers
Arm/Group | Be Well Care Well | Control
Number analyzed (Participants) | 115 | 67
units on a scale | 39.14 (5.21) | 41.51 (3.69)

3. Other Pre Specified Outcome: Change in Score on the Lifestyle Questionnaire
Description: The lifestyle questionnaire measured health and functioning. The physical activity subscale was used in this study, which had 18 items and ranged from 0-4 with higher scores representing more physical activity.
Time Frame: Baseline and 1-year follow-up
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Score on the Early Childhood Job Satisfaction Survey
Description: The Early Childhood Job Satisfaction Survey measures work satisfaction regarding co-worker relations, supervisor support, nature of the work itself, working conditions, and pay and promotion opportunities. The total score is used in this study and contains 55 items that range from 1-5. Higher scores on this scale represent higher job satisfaction.
Time Frame: Baseline and 1-year follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no adverse events in the current study
Groups:
- Be Well Care Well: There were no adverse events reported in the Be Well Care Well group.
- Control: There were not adverse events reported in the control group.
Arm/Group | Be Well Care Well | Control
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/67
Other Adverse Events (participants affected / at risk) | 0/115 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05310201/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT05310201/ICF_001.pdf